CLINICAL TRIAL: NCT06730152
Title: Efficacy of a WeChat Public Account-based Intervention for Smartphone Addiction Among Chinese Undergraduate Students: a Randomized Controlled Trial
Brief Title: WeChat Intervention for Smartphone Addiction in College Students: a Randomized Trial
Acronym: smartphone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Guifang Jin, Master's Degree Student, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 83244555; No.81973064 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-07

CONDITIONS: Smartphone Addiction
Keywords: smartphone addiction; behavior change; Information-Motivation-Behavioral Skills Model
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WeChat Information-Motivation-Behavioral Skills Model Intervention Group (Experimental): The intervention group would undergo a six-week intervention program. Researchers promoted a public WeChat account to the intervention group, and participants received the intervention by following the account. They automatically received pushed articles or videos, providing them with relevant knowledge about overcoming smartphone addiction. Furthermore, they would be motivated to quit their addiction through real-life cases of smartphone addiction etc., in addition to some practical skills of overcoming.
  Interventions: Behavioral: WeChat Intervention Based on the IMB Model
- Control group (No Intervention): without any intervention, maintain normal life and study state

INTERVENTIONS:
Behavioral: WeChat Intervention Based on the IMB Model — The intervention group would undergo a six-week intervention program. Researchers promoted a public WeChat account to the intervention group, and participants received the intervention by following the account. They automatically received pushed articles or videos, providing them with relevant knowledge about overcoming smartphone addiction. Furthermore, they would be motivated to quit their addiction through real-life cases of smartphone addiction etc., in addition to some practical skills of overcoming.
  Arms: WeChat Information-Motivation-Behavioral Skills Model Intervention Group

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of an intervention based on the Information-Motivation-Behavioral Skills (IMB) model to treat smartphone addiction in college students. The main questions it aims to answer are:

Does the IMB model-based intervention via WeChat public accounts significantly reduce smartphone addiction scores compared to a control group? Does the intervention lead to an increase in motivation and behavioral skills scores among participants? Researchers will compare the intervention group, which receives IMB-enhanced content through WeChat public accounts, to the control group, which maintains regular activities, to see if there are significant improvements in addiction scores, motivation, and behavioral skills in the intervention group.

Participants will:

Be stratified by gender and randomly assigned to either the intervention or control group.

The intervention group will receive information, motivation, and behavioral skills enhancement via WeChat public accounts over a period of 6 weeks.

Both groups will be assessed for smartphone addiction scores, information-motivation-behavioral skills scores, average daily smartphone use time, sleep duration, sleep quality, and somatic and psychological symptoms before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Meeting the criteria of the Smartphone Addiction Scale-Short Version (SAS-SV), with a score of ≥31 for males and ≥33 for females indicating smartphone addiction.

College students over 18 years old. Active use of WeChat software. Voluntary participation in this study and signing of the informed consent form.

Exclusion Criteria:

Currently not enrolled in school due to reasons such as suspension. Currently participating in other research projects. Self-reported diagnosis of any neurological or psychiatric disorder.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
smartphone addiction scale scores | From enrollment to the end of treatment at 6 weeks]
  Smartphone Addiction Scale: The Chinese version of the Smartphone Addiction Scale - Short Version (SAS-SV), containing 10 items. Minimum score of 6, Maximum score of 60, higher scores indicate more severe smartphone addiction .

SECONDARY OUTCOMES:
average daily smartphone use time | From enrollment to the end of treatment at 6 weeks
  assessed as, "Average daily cell phone use in the last month."
sleep duration | From enrollment to the end of treatment at 6 weeks]
  assessed as, "Actual sleep time per night for the last 1 month."
sleep quality | From enrollment to the end of treatment at 6 weeks]
  assessed as, "How would you rate your sleep quality in the past month

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon M, Lee JY, Won WY, Park JW, Min JA, Hahn C, Gu X, Choi JH, Kim DJ. Development and validation of a smartphone addiction scale (SAS). PLoS One. 2013;8(2):e56936. doi: 10.1371/journal.pone.0056936. Epub 2013 Feb 27. PMID 23468893
- [Background] Bi J, Yang W, Hao P, Zhao Y, Wei D, Sun Y, Lin Y, Sun M, Chen X, Luo X, Li S, Zhang W, Wang X. WeChat as a Platform for Baduanjin Intervention in Patients With Stable Chronic Obstructive Pulmonary Disease in China: Retrospective Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 2;9(2):e23548. doi: 10.2196/23548. PMID 33528369
- [Background] Bakir E, Cavusoglu H, Mengen E. Effects of the Information-Motivation-Behavioral Skills Model on Metabolic Control of Adolescents with Type 1 Diabetes in Turkey: Randomized Controlled Study. J Pediatr Nurs. 2021 May-Jun;58:e19-e27. doi: 10.1016/j.pedn.2020.11.019. Epub 2020 Dec 25. PMID 33371976